CLINICAL TRIAL: NCT00815230
Title: Effect of Cardiac Computed Tomography Angiography on the Blood Reactive Oxygen Species Level
Status: Withdrawn | Type: Observational
Why Stopped: because of unexpected administrative barrier, it was very difficult to enroll case.
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Zei-Shung Huang, associate professor, Department of Internal Medicine, NTUH, National Taiwan University Hospital
Other Study IDs: 200812057R
Record Dates: First submitted 2008-12-25; First posted 2008-12-29 (Estimated); Last update posted 2009-05-19 (Estimated); Status verified 2008-12

CONDITIONS: Radiation Injury
Keywords: radiation injury; computed tomography; reactive oxygen species; free radicals
MeSH Terms: conditions — Radiation Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — only peripheral blood will be collected for measurement of reactive oxygen species.
Oversight: Data Monitoring Committee: No

SUMMARY:
The clinically widely used X-ray computed tomography examination has a low-grade radiation effect and recently has attracted much attention concerning the possible adverse effects of radiation on human body [ref. 1-5]. The radiation is harmful to human tissues and cells mainly because it can interact with water (which makes up to 80% of cells) to generate reactive oxygen species (ROS), especially the formation of hydroxyl radicals. So far as we can reach, there is no report concerning the relation between X-ray computed tomography examination and the blood ROS level. Therefore, we wish to conduct this study to clarify if the cardiac computed tomography angiography (cardiac CTA) may induce a higher level of ROS in the peripheral blood.

Study subjects will be OPD patients who are arranged for cardiac CTA examination because of suspect coronary artery disease (CAD). In total, twenty cases will be enrolled for the study. The formal consent will be delivered and explained to the patients and families after the arrangement of cardiac CTA. It then will be retrieved just before the performance of cardiac CTA.

For each enrolled case, peripheral blood will be sampled three times (once before and twice after the performance of cardiac CTA). Totally 60 blood samples will be collected from 20 study subjects within 3 months (January 1 ~ March 31, 2009). ROS level in the collected blood samples will be then measured, compared, and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* subjects who are arranged for cardiac CTA examination because of suspect coronary artery disease.

Exclusion Criteria:

* none

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study subjects will be OPD patients who are arranged for cardiac CTA examination because of suspect coronary artery disease.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2009-01; Study Completion 2009-03 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- NTUH, Taipei, Taiwan